CLINICAL TRIAL: NCT02348567
Title: Unannounced or Announced Periodic Hospital Surveys: A Study Protocol for a Nationwide Cluster-randomised, Controlled Trial
Brief Title: Unannounced Periodic Surveys on Public Hospitals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Danish Center for Healthcare Improvement (Other)
Collaborators: Institute for Quality and Accreditation in Healthcare (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1234; 12345 (Other: Danish Center for Healthcare Improvements)
Record Dates: First submitted 2014-09-15; First posted 2015-01-28 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Accreditation
Keywords: Health care, accreditation, unannounced survey, cluster randomized controlled trial, quality improvement, organisational development
MeSH Terms: interventions — Patient Safety

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- announced hospital surveys (Active Comparator): Eleven hospitals will receive announced surveys (control group)
  Interventions: Other: announced hospital surveys
- unannounced hospital surveys (Experimental): 12 hospitals will receive unannounced surveys (intervention group).
  Interventions: Other: Unannounced hospital surveys

INTERVENTIONS:
Other: Unannounced hospital surveys — This is a cluster-randomised controlled trial performed at hospital level. We hypothesise that unannounced surveys produce less successful assessments of patient safety compared to announced surveys (conventional/control). This study defines less successful as less compliance with the included standards and performance indicators.
  Other Names: quality development, patient safety
  Arms: unannounced hospital surveys
Other: announced hospital surveys
  Arms: announced hospital surveys

SUMMARY:
Introduction: Accreditation programmes for healthcare systems have been implemented in more than 70 countries to stimulate high-quality organisational performance. Several Danish healthcare institutions are covered by the Danish Healthcare Quality Programme (DDKM) and all Danish public hospitals have been accredited according to the DDKM since 2010.

The dates of each survey are currently being announced 8-10 months beforehand. Announcing surveys has been criticised for creating an "arranged reality". It has therefore been suggested that a national intervention be conducted to evaluate the effect of unannounced hospital surveys.

Methods and analysis: All public somatic and psychiatric hospitals in Denmark (n=30) were invited to participate in the trial. Twenty-three hospitals (77%) (3 university hospitals, 5 psychiatric hospitals, and 15 general hospitals) agreed to participate and to be randomised to one of the trial clusters. Eleven hospitals will receive announced surveys (control group) and 12 hospitals will receive unannounced surveys (intervention group).We hypothesise that hospitals receiving unannounced surveys will be rated as less successful than hospitals receiving announced surveys, defined as meeting less compliance with accreditation standards and performance indicators. Nine experienced surveyors employed and educated by The Danish Institute for Quality and Accreditation in Health Care (IKAS) will be responsible for conducting the surveys according to an abbreviated version of the current Danish periodic survey. The outcome is compliance with indicators reflecting organisational performance. Compliance will be analysed using logistic or linear regression analysis with random effects, contingency tables, and Pearson's chi-squared test or Fishers exact test, whichever is most appropriate.

Ethics and Dissemination: This trial is pending ethics approval from Research Ethichs Comite for North Denmark Region. The findings from this randomised controlled trial will be disseminated through peer-reviewed journals, national and international conferences and will be utilised as health care political decision making for the future national accreditation programme. In addition, the results will facilitate to validate the effect of unannounced hospital surveys; given the issues of currently meeting an "arranged reality" during hospital surveys, this seems extremely desirable.

DETAILED DESCRIPTION:
Accreditation by external audit to validate that healthcare organisations' operations and practices satisfy agreed high-quality service criteria are being conducted in more than 70 countries (1,2). In 2003, the Danish government and The Danish Regions (responsible for all public hospitals) decided to implement a nationwide model of quality in healthcare which involves formal accreditation of all Danish public hospitals. In 2007, a national Institute for Quality and Accreditation in Healthcare (IKAS) was formed to develop The Danish Healthcare Quality Programme (DDKM); and since 2010, all public hospitals have been accredited based on announced on-site surveys which are conducted every third year (including a periodic midterm survey). Other types of healthcare institutions are now also included in the program and accredited on a regular basis (e.g. private hospitals covered by the extended free hospital choice, pharmacies, and nursing homes), and a plan for accreditation in general practices is currently (2014) being negotiated (3-5).

The DDKM is based on announced surveys and the procedure of pre-announcing the dates for all surveys has been criticised for creating an "arranged reality" and for not reflecting the daily work with quality of care. This criticism is not unique to the Danish setting, but has been raised in a number of countries that operate accreditation systems based upon announced surveys (6,7). Another possible negative effect of announcing the surveys is the considerable amount of time and human resources that are used to prepare for the announced survey which implies that less time is available for patient care in the period of preparations (6). It has been proposed that unannounced accreditation surveys may be instrumental in alleviating these problems. An unannounced survey is an external visit paid to an organisation without prior notice of when the visit will take place (2).

Unannounced surveys have been used for several years by The Joint Commission in the United States and the Aged Care Standards and Accreditation Agency in Australia, but to our knowledge no peer-reviewed literature has been published on the experiences of changing the procedure from announced to unannounced surveys (2,7,8). Only one project, launched by The Centre for Clinical Governance Research (CCGR) in Australia in 2012, encompasses an empirical test of short-notice surveys in two accreditation programmes. This study was conducted in a paired design where short-notice surveys are compared with the most recent and most advanced notification survey. The study found that use of the short-notice survey approach to the rating of organisational performance was less successful than the advanced notification survey (5% significance level, P=0.044) (9).

The present trial is designed by IKAS and the Danish Center for Healthcare Improvements (DCHI) to inform a decision whether or not to implement unannounced accreditation surveys in the 3rd version of the DDKM in 2016. In September 2013, the IKAS Board of Directors decided to approve and finance the project, and it is expected that the results from the present trial will be available for the Board's decision in 2015.

To provide the best possible basis for political decision-making, the present study is designed as a nationwide cluster-randomised, controlled trial including general hospitals, university hospitals, and psychiatric hospitals from all five regions in Denmark. The objective of this trial is to evaluate the effect of unannounced hospital surveys based on findings of a survey embracing an abbreviated set of the national accreditation standards and performance indicators from the DDKM version 2. We hypothesise that unannounced surveys produce less successful measures of organisational performance than announced surveys. This study defines less successful as less compliance with the included standards and performance indicators.

ELIGIBILITY:
Inclusion Criteria:

public hospitals:

* psychiatric hospitals
* university hospitals
* general hospitals

Exclusion Criteria:

* private hospitals

NOTE: "accept of healthy volunteers": we assess accreditation indicators at hospital level. human subjects (hospital staff and patients) are interviewed in relation to hospital accreditation indicators performed by hospital surveyors.

Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
hospital accreditation standards/indicators | 25 weeks
  The surveyors will classify each assessed performance indicator (n=113) in predetermined phrases that covers the organisational performance. Each phrase is assigned a level of performance (1-4), to enable a convertion of data into categorical ordinal variables. The predetermined phrases are determined as; "consistent implementation"=1, "consistent implementation with single deviations"=2, "weak implementation"=3, and "missing implementation"=4. All findings will be accumulated on each performance indicator.

CONTACTS AND LOCATIONS:
Overall Officials: Lars H Ehlers, Professor, Study Director — Danish Center for Healthcare Improvement
Locations (1):
- Danish Center for Healthcare Improvements, Aalborg, Denmark

REFERENCES:
- [Background] Greenfield D, Moldovan M, Westbrook M, Jones D, Low L, Johnston B, Clark S, Banks M, Pawsey M, Hinchcliff R, Westbrook J, Braithwaite J. An empirical test of short notice surveys in two accreditation programmes. Int J Qual Health Care. 2012 Feb;24(1):65-71. doi: 10.1093/intqhc/mzr074. Epub 2011 Dec 2. PMID 22140191
- [Derived] Ehlers LH, Simonsen KB, Jensen MB, Rasmussen GS, Olesen AV. Unannounced versus announced hospital surveys: a nationwide cluster-randomized controlled trial. Int J Qual Health Care. 2017 Jun 1;29(3):406-411. doi: 10.1093/intqhc/mzx039. PMID 28419255